CLINICAL TRIAL: NCT06670846
Title: Management of Preoperative Anxiety in Children: Could a Lollipop Be the Solution?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Mehdi Trifa, Head of the anesthésia and intensive care department, Tunis University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 302023
Record Dates: First submitted 2024-10-21; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Anxiety, Preoperative
Keywords: anxiety; children; anesthesia; distraction; midazolam
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Chidren were randomized into two groups to receive either intranasal midazolam at 0.3 mg/kg (group M) or distraction using a lollipop (group L) 15 minutes before entering the operating room
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lollipop arm (Experimental): Distraction using a lollipop (group L) 15 minutes before entering the operating room
  Interventions: Device: Lollipop
- Midazolam arm (Active Comparator): Intranasal midazolam at 0.3 mg/kg 15 minutes before anesthesia
  Interventions: Drug: distraction using intranasal Midazolam

INTERVENTIONS:
Device: Lollipop — Distraction using a Lollipop 15 minutes before anesthesia
  Arms: Lollipop arm
Drug: distraction using intranasal Midazolam — Distraction using intranasal Midazolam 15 minutes before anesthesia
  Arms: Midazolam arm

SUMMARY:
The aim of the study is to evaluate the effectiveness of distraction using a lollipop versus premedication with intranasal midazolam to manage preoperative anxiety in pediatric anesthesia.

DETAILED DESCRIPTION:
Participants were randomized into two groups to receive either intranasal midazolam at 0.3 mg/kg (group M) or distraction using a lollipop (group L) 15 minutes before entering the operating room. The anesthetic technique was standardized: a peripheral intravenous line, intravenous induction (propofol and fentanyl), airway management with an age-appropriate IGEL mask, and maintenance with sevoflurane. Anxiety was assessed using the modified Yale Preoperative Anxiety Scale (mYPAS) before and after premedication. The investigators also evaluate the level of sedation upon entering the operating room, the quality of parent separation, acceptance of the facemask during induction, and emergence of agitation using the Pediatric Anesthesia Emergence Delirium Scale (PAEDS).

ELIGIBILITY:
Inclusion Criteria:

* Age > 4 ans , ASA 1 ou 2

Exclusion Criteria:

* Children who rejected premedication - The occurrence of perioperative complications

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 63 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
anxiety | immediatly before premedication and 15 minutes after premedication
  Anxiety was assessed using the modified Yale Preoperative Anxiety Scale (mYPAS) before and after premedication. The myPAS score includes 5 items, with a minimum value of 4 and a maximum value of 22; a higher score indicates a major anxiety.

SECONDARY OUTCOMES:
agitation | 10 minutes after extubation
  Emergence agitation assessed using the Pediatric Anesthesia Emergence Delirium Scale (PAEDS), which has a minimum score of 0 and a maximum score of 20. A higher score indicates more severe agitation during emergence from anesthesia.
parent separation | 15 minutes after premedication
  The quality of parent separation Defined by 3 items: the child waits near their parents rated as 1, clings to their parents rated as 2, or refuses separation rated as 3

CONTACTS AND LOCATIONS:
Locations (1):
- Bechir Hamza hospital, Tunis, Tunis Governorate, Tunisia